CLINICAL TRIAL: NCT00503256
Title: Genetic Study of Chronic Lymphocytic Leukemia Families
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ID03-0117
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; Lymphoma; Questionnaire; Survey; CLL
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cheek cell sample collection that will be used for special tests to look for genes that may play a role in the development of CLL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLL - Linkage Families: Gene identification related to Chronic lymphocytic leukemia (CLL) development
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires each taking 60 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this research is to identify genes that may be related to the risk of developing CLL.

Objectives:

The objective of this study to investigate possible candidate susceptibility genes for familial chronic lymphocytic leukemia (CLL) by identifying and recruiting high-risk families. Through our ongoing study of familial aggregation in CLL kindreds (protocol 2003-0498 'Genetic Study of Chronic Lymphocytic Leukemia'), we have identified CLL patients who have one or more living or dead relative(s) affected with CLL or other leukemias or lymphomas. We will also identify patients in high-risk families from referrals from leukemia clinicians and from self-referrals from patients who learn about our study from the ClinicalTrials.gov website. We plan to invite probands (patients diagnosed with CLL) and their family members with other leukemias and lymphomas and a sample of unaffected relatives to participate in a genetic/linkage study. We will obtain demographic and clinical information along with specimens (blood or buccal samples) from all participants. These families will be part of the Genetic Epidemiology of CLL Consortium, a multicenter, multidisciplinary consortium, based at the Mayo Clinic Cancer Center under the direction of Susan Slager, PhD. This is funded from NCI through a subcontract with Mayo Clinic.

Genotypic data will be analyzed at Mayo Clinic, and coded, de-identified data will be shared with the NIH Genome-Wide Association Studies (GWAS) data repository.

DETAILED DESCRIPTION:
This study does not involve taking any medications.

You will be asked to provide study personnel with authorization to request medical records from your physician, the hospital, and/or from other health care facilities where you were diagnosed with cancer. The information gathered will be used to help verify the diagnosis. Study personnel may also need to contact you in the future by phone, mail, or e-mail in order to ask questions about the status of your health.

For this research study, you will be asked to have around 4 tablespoons of blood drawn from a vein in your arm or you will also be asked to provide a sample of cheek cells by spitting into a collection container. The blood and cheek cell samples will be used for special tests to look for genes that may play a role in the development of CLL. You will also be asked to complete a family history questionnaire and a risk factor questionnaire. The family history questionnaire and the risk factor questionnaire will each take 60 minutes to complete. You will need to contact your family members before you send the completed family history questionnaire back to the study staff. You must ask for their permission to send the study staff their contact information. Family members with CLL or other leukemias or lymphomas, as well as a sample of your unaffected family members, will then be contacted by study personnel about participating in the study.

If you live in Houston, or the surrounding area, study personnel can arrange to collect the samples at the time and place of your convenience. If you do not live in the Houston area, sample collection instructions and supplies will be mailed to you. The blood sample may be drawn at your doctor's office, or at a clinic or hospital of your choice. All mailing costs will be paid by the study. No travel to M. D. Anderson will be required.

All blood and cheek cells collected will only be used by researchers involved in this study. Genetic information from the analysis of your blood and cheek cells will be included in a repository of genetic information at the National Institutes of Health, but no personal identifying information will be sent. All information will be kept confidential. Neither you nor your doctor will receive the results of these tests and they will NOT be put in your medical record.

This is an investigational study. Up to 450 participants will be enrolled by M. D. Anderson researchers. A total of 4000 participants will be enrolled in this multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CLL who have living or dead relatives affected with CLL. They must agree to complete a risk factor questionnaire and a family history questionnaire, and to donate a 50mL blood specimen or a buccal specimen.
2. Relatives of the CLL patients who have CLL or other lymphoproliferative disorders (i.e., leukemia & lymphoma). They must agree to complete a risk factor questionnaire and donate a 50mL blood specimen or a buccal specimen. They will need to sign an authorization to release their medical records so that we can confirm their diagnosis.
3. A sample of unaffected relatives of the CLL patients. They must agree to complete a risk factor questionnaire and donate a 50mL blood specimen or a buccal specimen.

Exclusion Criteria:

1) No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with chronic lymphocytic leukemia (CLL) and their living unaffected or affected relatives.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2003-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Candidate susceptibility genes for familial chronic lymphocytic leukemia (CLL) | Data collection over 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, BS, Principal Investigator — M.D. Anderson Cancer Center; Susan Slager, Ph.D., Study Director — Mayo Clinic
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org